CLINICAL TRIAL: NCT05845580
Title: The Patient Autonomy and Statin Therapy Adherence (PASTA) Trial: A Randomized Controlled Trial Comparing Adherence to Atorvastatin Therapy in Primary Prevention Patients Who Decline Statin Therapy, When Given a Choice Between Atorvastatin and Red Yeast Rice Extract as Their Initial Therapy
Brief Title: Patient Autonomy and Statin Therapy Adherence
Acronym: PASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Minneapolis Heart Institute (Other); Kreiskrankenhaus Rotenburg an der fluda (Unknown); Klaipėda University (Other)
Responsible Party: Principal Investigator, Ali Aldujeli, Cardiovascular disease consultant, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUHSKC-204
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Drug Adherence
Keywords: Statins; Patient autonomy; Red yeast rice extract; Patient-centered care; Primary prevention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to receive either atorvastatin therapy or red yeast rice extract and then atorvastatin. The two arms will be run concurrently, and patients in each arm will be assessed for adherence and outcomes over the same period of time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient centered care (Experimental): Patients concern of refusing statin therapy will initially be addressed.
  Interventions: Other: Red yeast rice extract initial therapy followed later on by statin therapy
- Guideline-centered care (Active Comparator): patients will be prescribed the standard of care regardless of their concerns toward statin therapy.
  Interventions: Other: Statin therapy

INTERVENTIONS:
Other: Red yeast rice extract initial therapy followed later on by statin therapy — Patients will be offered red yeast rice extract to achieve a target LDL-cholesterol level of <2.6 mmol/L, as recommended by the 2019 ESC/EAS guidelines. If a patient's LDL-cholesterol level remains above the target during follow-up, they will be informed that the natural alternative was ineffective, and they will be prescribed atorvastatin.
  Arms: Patient centered care
Other: Statin therapy — Patients will be provided reassurance through a short, semi-structured discussion on the excellent safety profile of statins, similar to a typical interaction between a clinician and patient. They will then be prescribed atorvastatin.
  Arms: Guideline-centered care

SUMMARY:
The rationale for the Patient Autonomy and Statin Therapy Adherence (PASTA) trial is based on the fact that statin therapy is a highly effective and evidence-based treatment for reducing the risk of cardiovascular disease. However, despite the proven benefits of statin therapy, a significant proportion of patients decline to take statins due to concerns about side effects, safety, or a preference for alternative treatments.

One potential strategy to improve statin adherence in patients who decline therapy is to give patients more autonomy in selecting their treatment options. By offering patients a choice between a traditional statin medication (atorvastatin) or a "natural" statin alternative (red yeast rice extract) and involving them in the goal-setting process for their LDL-C levels, patients may feel more empowered and engaged in their own care.

The PASTA trial aims to evaluate whether greater patient autonomy leads to improved adherence to statin therapy in patients who decline initial therapy. By measuring the impact of patient autonomy on statin adherence, the study results may provide valuable insights into how to improve patient engagement and health outcomes in a population that may be hesitant to initiate statin therapy.

DETAILED DESCRIPTION:
Statin therapy is an integral tool in the primary and secondary prevention of atherosclerotic cardiovascular disease (ASCVD). Higher compliance with their statin therapy is associated with a lower risk of mortality in a step-wise manner . Despite this, rates of statin compliance are abysmally low. Prior studies suggest that less than 40% of primary prevention patients are compliant with their prescribed statin therapy. Individuals who have suffered a prior MI have an incremental improvement in compliance to around 60%. Younger individuals and women appear to have exceptionally low rates of compliance to statin therapy . Low rates of compliance remains a significant barrier to reducing the burden of ASCVD, with some suggesting efforts to increase compliance can have an oversized impact on reducing rates of ASCVD .

On the other hand, patients often prefer "natural" therapies over conventional medicine for a variety of reasons. Monacolin-K is a naturally occurring molecule in red yeast-rice extract, a commonly used health supplement. It is structurally identical to lovastatin and has been shown to reduce LDL-C levels and ASCVD events in randomized placebo controlled trials.

Patient autonomy is a core bioethical principle affirming the right of the patient to determine the trajectory of their health care at times. This bioethical principle has been referred to as "first among equals", implying that it is the most important bioethical principle. The role of autonomy in patient compliance is not entirely clear, but there is evidence that suggests that increased patient autonomy in the decision-making process can result in higher rates of long term compliance.

ELIGIBILITY:
Inclusion criteria

1. Moderate atherosclerotic cardiovascular disease risk
2. Decline statin therapy

Exclusion criteria

1. Dementia
2. Severe Mental Illness
3. History of statin intolerance
4. High-risk for atherosclerotic cardiovascular disease
5. Currently on lipid lowering therapy
6. Currently taking red yeast rice extract
7. Pregnant or breast feeding
8. Concomitant use of the following drugs: anti-retroviral therapy, niacin, calcineurin inhibitors, mTOR inhibitors, amiodarone, and fibrates

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of statin compliance | 8 months
  Based on pharmacy refill records. Values per patient can range from 0-6 according to the number of refills.

SECONDARY OUTCOMES:
Rate of perceived side-effects from statin use | 8 months
  including muscle aches, fatigue, mental fog, and gastrointestinal upset.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05845580/Prot_000.pdf